CLINICAL TRIAL: NCT06313541
Title: A Multicenter, Randomized Controlled Clinical Trial of Treatment Response Adapted Hybrid Radiotherapy in Metastatic Non-small Cell Lung Cancer Receiving First-line Immunotherapy
Brief Title: Treatment Response Adapted Hybrid Radiotherapy in Metastatic Non-small Cell Lung Cancer Receiving First-line Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-Lung-LDRT/SBRT
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Platinum Compounds

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1/PD-L1 inhibitor combined with chemotherapy (Active Comparator)
  Interventions: Drug: PD-1/PD-L1 inhibitor combined with platinum-based chemotherapy
- Treatment response adapted hybrid radiotherapy plus PD-1/PD-L1 inhibitor and chemotherapy (Experimental)
  Interventions: Radiation: SBRT or LDRT; Drug: PD-1/PD-L1 inhibitor combined with platinum-based chemotherapy

INTERVENTIONS:
Radiation: SBRT or LDRT — Radiotherapy: (1) Low dose radiotherapy (LDRT) : a dose of 2 Gy/1 Fx was given to all visible lesions in the whole body within 1 week before the first course of PD-1/PD-L1 inhibitor combined with chemotherapy (different parts of the lesion could be irradiated separately, but it was required to be completed within 1 week); (2) SBRT: patients received first-line immunotherapy combined with chemotherapy, and their response was evaluated every 6 weeks. Individualized SBRT was planned based on the treatment responses.
  Arms: Treatment response adapted hybrid radiotherapy plus PD-1/PD-L1 inhibitor and chemotherapy
Drug: PD-1/PD-L1 inhibitor combined with platinum-based chemotherapy — The control group received standard PD-1/PD-L1 inhibitor combined with platinum-based chemotherapy as first-line treatment, and the experimental group received extra treatment response adapted hybrid radiotherapy.

SUMMARY:
This study is a multicenter, randomized controlled clinical trial to explore the preliminary efficacy and safety of treatment response adapted hybrid radiotherapy (LDRT and SBRT) in the first-line treatment of immunotherapy combined with chemotherapy for advanced driver-gene negative NSCLC, and to provide new ideas for the comprehensive treatment of advanced NSCLC

ELIGIBILITY:
Inclusion Criteria:

* ECOG functional status score was 0-1.
* Histologically confirmed stage IV primary NSCLC;
* Genetic testing showed that the common driver genes including EGFR, ALK and ROS-1 were negative;
* Patients with brain metastases were eligible if they were neurologically asymptomatic and had stable disease without receiving systemic glucocorticoids;
* According to the investigator's judgment, the patient does not need to receive palliative radiotherapy for any site at present;
* Male/female of childbearing age agreed to use contraception (surgical ligation or oral contraceptive/intrauterine device plus condom) during the trial;
* Life expectancy ≥3 months;
* One week before enrollment, the organ function level met the following criteria:

  ① Bone marrow function: hemoglobin ≥80g/L, white blood cell count ≥4.0*10^9/L or neutrophil count ≥1.5*10^9/L, platelet count ≥100*10^9/L;

  ② Liver: serum total bilirubin level ≤1.5 times upper limit of normal, direct bilirubin level must be ≤1.5 times upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times upper limit of normal;

  ③ Kidney: serum creatinine < 1.5 times upper limit of normal or creatinine clearance ≥50ml/min, urea nitrogen ≤200mg/L; Serum albumin ≥30g/L;
* Patients must be able to understand and voluntarily sign the informed consent form.

Exclusion Criteria:

* The patient had severe autoimmune diseases: active inflammatory bowel disease (including Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (such as Wegener's granulomatosis), etc.
* Symptomatic interstitial lung disease or active infectious/non-infectious pneumonia;
* Patients with risk factors for intestinal perforation: active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal cancer, or other known risk factors for intestinal perforation;
* History of other malignant tumors;
* Patients with active infection, heart failure, myocardial infarction, unstable angina or unstable arrhythmia within the past 6 months;
* Medical examination or clinical findings, or other uncontrollable conditions that the investigator considers may interfere with the results or increase the patient's risk of treatment complications;
* Patients who were considered by the investigator to have lesions requiring palliative and subtractive radiotherapy;
* Mixed with small cell lung cancer components;
* Lactating or pregnant women;
* Congenital or acquired immunodeficiency diseases including human immunodeficiency virus (HIV), organ transplantation or allogeneic stem cell transplantation;
* Known HBV, HCV, active pulmonary tuberculosis infection;
* Patients had received a cancer vaccine or received another vaccine within 4 weeks before starting treatment (note: injectable seasonal influenza vaccine is usually inactivated, so vaccination is allowed, while intranasal vaccine is usually live attenuated, so it is not allowed);
* Patients with concurrent use of other immune agents, chemotherapy drugs, drugs in other clinical studies, and long-term use of cortisol were excluded.
* Patients with mental disorders, substance abuse, or social problems that affect adherence were excluded from the study after physician review;
* Patients who are allergic to or contraindicated to PD-1 monoclonal antibody or chemotherapy drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Two years
  The time from enrollment to disease progression or death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.

SECONDARY OUTCOMES:
Overall Survival | Two years
  The time from enrollment to death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
Objective response rate | Two years
  According to RECISIT1.1 criteria, the proportion of patients achieving CR and PR as their best response before initial disease progression was evaluated.
Progression free survival 2 | Two years
  The time between enrollment and the observation of second disease progression or the occurrence of death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
Treatment-related adverse event | Two years
  Investigator-assessed treatment-related adverse events were recorded and assessed according to CTCAE5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China